CLINICAL TRIAL: NCT04320485
Title: Evaluation of the Clinical Specificity of the Active Anthrax Detect™ Plus (AAD Plus) Lateral Flow Immunoassay (LFI)
Status: Completed | Type: Observational
Sponsor: InBios International, Inc. (Industry)
Collaborators: Fast-Track Drugs & Biologics, LLC (Unknown); Biomedical Advanced Research and Development Authority (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: AAD Plus-2018-01
Record Dates: First submitted 2020-03-22; First posted 2020-03-25 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Anthrax
Keywords: Anthrax; Lateral flow immunoassay; Diagnostics
MeSH Terms: conditions — Anthrax

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 8 milliliters of blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

INTERVENTIONS:
Diagnostic Test: Active Anthrax Detect™ Plus (AAD Plus) — A lateral flow immunoassay rapid test (AAD Plus) for early and presumptive diagnosis of inhalational anthrax.

SUMMARY:
The primary objective of the study is to determine the estimated clinical specificity of the AAD Plus. A secondary objective is to determine the estimated sensitivity of the AAD Plus as 10% of the study subject samples will be contrived to be positive.

DETAILED DESCRIPTION:
This study is a multi-site trial assessing the clinical specificity of AAD Plus using capillary blood, venous blood, and venous serum samples collected from presumptive anthrax negative subjects who present with symptoms consistent with cold, flu or other bronchial and febrile infections in the US. At least 440 subjects who meet the study eligibility criteria will have 3 blood samples from a single time point tested with the AAD Plus device. The samples will be: 1) capillary blood collected by finger stick; 2) venous blood collected in a sodium citrate anticoagulant tube; and, 3) serum obtained from venous blood collected in a serum separator tube. The capillary blood sample will be tested immediately to avoid clotting by an unblinded staff member. The venous blood and serum samples will be tested by a blinded staff member as soon as possible after preparation. Additional aliquots of the serum sample will be prepared and stored frozen at -20 ± 2°C or colder for possible additional reference testing [CDC reverse-transcriptase polymerase chain reaction (RT-PCR) assay (K140426)] in the event that any of the subject's capillary blood, venous blood, or serum sample is positive.

At each clinical site, subjects' paired venous whole blood and serum samples will be randomly selected such that 10% of all subjects' samples (total of 40) will be spiked with recombinant anthrax lethal factor (LF) to prepare a contrived positive sample. Each clinical site will be provided a unique randomization list by the Data Management Center that identifies, which subjects will be randomized for spiking with LF. The numbers of spiked samples will be distributed approximately equally between all sites. An unblinded site staff member will prepare the blinded, spiked (from 40 subjects selected for spiking) and unspiked (from 400 subjects that are not selected for spiking) venous blood and serum specimens to be tested by a blinded staff member. Before the venous blood sample and serum specimens (from subjects selected for spiking) are spiked; the unblinded staff member will also test all unspiked samples on the AAD Plus and record the results. Then the spiked venous blood and serum sample will be given to the blinded staff member for testing. Thus, blinded staff will receive whole blood and serum samples that could be either unspiked (presumed negative) or spiked (presumed positive) to preserve the blind. In the rare event that the AAD Plus test result is positive on the unspiked sample tested by the unblinded staff member, then the unblinded staff member will give the unspiked sample from this subject to the blinded operator for AAD Plus testing and the subject's serum sample will be sent for reference testing as described above. Blinded staff will remain blinded throughout the study to the contrived spiking of the whole blood and serum samples as to which samples were contrived.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18 to 90 years of age.
2. Current symptoms consistent with cold, flu or other bronchial and febrile infections. The subject must currently (day of consent) have at least one of the following symptoms: fever, chills, chest discomfort, shortness of breath, cough, dizziness/confusion, nausea, headache, sweats, fatigue, or body aches.

Exclusion Criteria:

1. Nursing home residents
2. Inmates/subjects in police custody
3. Unable to understand verbal or written language of the consent or require a Legal Authorized Representative for consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female subjects, 18 to 90 years of age, with symptoms consistent with cold, flu or other bronchial and febrile infections.
Sampling Method: Probability Sample
Enrollment: 450 (Actual)
Dates: Start 2020-03-25 (Actual); Primary Completion 2020-12-17 (Actual); Study Completion 2020-12-17 (Actual)

PRIMARY OUTCOMES:
The estimated specificity of the AAD Plus test. | Day of enrollment.
  For the estimated specificity, the negative percent agreement (NPA) will be calculated from testing unspiked specimens from 400 subjects (with presumed negative samples).

SECONDARY OUTCOMES:
The percent positive agreement (PPA) | Day of enrollment.
  The percent positive agreement (PPA) of the contrived serum specimens will be calculated under the assumption that all spiked specimens are true positives.

CONTACTS AND LOCATIONS:
Overall Officials: Marketa Hnilova, PhD, Study Director — InBios International
Locations (4):
- United States (4):
  - Fiel Family and Sports Medicine/CCT Research, Tempe, Arizona
  - Hometown Urgent Care and Research, Cincinnati, Ohio
  - Hometown Urgent Care and Research, Columbus, Ohio
  - Hometown Urgent Care and Research, Dayton, Ohio

IPD SHARING:
Plan to Share IPD: No